CLINICAL TRIAL: NCT00106600
Title: A Phase I/II Study of Pixantrone (BBR 2778) in Patients With Refractory Acute Myelogenous Leukemia (AML)
Brief Title: Pixantrone (BBR 2778) in Patients With Refractory Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIX109
Record Dates: First submitted 2005-03-28; First posted 2005-03-29 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2007-08

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

INTERVENTIONS:
Drug: Pixantrone IV infusion

SUMMARY:
The goal of this study is to find the safest dose of Pixantrone (BBR 2778) that can be given to patients with Acute Myelogenous Leukemia (AML). After the safest dose is found, up to an additional 86 patients will be enrolled. During this part of the study, the safety and effectiveness will be evaluated.

DETAILED DESCRIPTION:
This is an open label, single center, phase I/II study of pixantrone in patients with refractory AML. Pixantrone will be administered for three consecutive days on days 1, 2 and 3 of each 21-day cycle, for up to two cycles.

The study has 2 parts; phase I and phase II. In the phase I part of the study, the maximum tolerated dose (MTD) for pixantrone as a single agent in patients with refractory AML will be determined. In the phase II part of the study, up to an additional 86 patients will be treated at the MTD to assess disease response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with morphologically confirmed diagnosis of relapsed AML with French-American-British (FAB) classification other than M3. Relapse should be demonstrated by the presence of greater than 5% leukemic blasts in the bone marrow or reappearance of greater than 5% leukemic blasts in the peripheral blood within 14 days of registration.

Eligible patients include the following:

* Patients with secondary AML, including patients with prior myelodysplastic syndromes (MDS)
* Patients who were initially unresponsive to induction therapy
* Patients in first or second relapse from prior therapy or hematopoietic stem-cell transplant (HSCT)

  * A period of at least 21 days must have elapsed from the completion of prior chemotherapy (with or without anthracyclines) and investigational agents to the first dose of treatment in this study, and all acute toxicities from prior therapy must have resolved (with the exception of alopecia).
  * Age >/= 18 years of age, and able to give informed consent.
  * ECOG performance status of 0, 1 or 2.
  * Bilirubin < 1.5 x institution's upper limit of normal (ULN), AST and ALT < 1.5 x institution's ULN, creatinine < 2 mg/dL.
  * LVEF >/= 50% as measured by MUGA scan or 2-D ECHO within 14 days prior to registration. Either method is acceptable for measuring LVEF; however, the same method must be used throughout treatment and follow-up.
  * Patients (male or female) of reproductive potential must commit to use adequate contraception (as defined by the investigator) during study treatment and for 6 months after the last day of study drug administration.
  * Patients must have signed an approved informed consent prior to beginning protocol specific procedures

Exclusion Criteria:

* Prior treatment with a cumulative dose of doxorubicin or equivalent exceeding 450 mg/m2 according to the following calculation index: X/450 + Y/160 < 1 where X is the doxorubicin dose in mg/m2 and Y is the mitoxantrone dose in mg/m2.
* Clinical or documented central nervous system (CNS) involvement with AML.
* Any uncontrolled active infection that requires antibiotics.
* History of Human Immunodeficiency Virus (HIV).
* Acute hepatitis, or known chronic hepatitis.
* Unstable cardiovascular conditions, including: cardiac arrhythmias, angina, or myocardial infarction within the past 6 months.
* Pregnant women or nursing mothers.
* Prior malignancy except: curatively treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in remission, or any other cancer from which the patient has been disease-free for 5 years.
* Any condition which, in the judgment of the investigator, would place the patient at undue risk, interfere with the results of the study, or make the patient otherwise unsuitable.
* Any circumstance at the time of study entry that would preclude completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Phase I: To determine the maximum tolerated dose (MTD) of Pixantrone (BBR 2778) in patients with refractory acute myelogenous leukemia (AML)
Phase II: To evaluate the activity of pixantrone in this patient population in terms of objective responses

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States